CLINICAL TRIAL: NCT01705899
Title: Islet Allotransplantation in Type 1 Diabetes
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Pausing of allotransplant program due to logistic issues.
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2006H0200
Record Dates: First submitted 2012-05-03; First posted 2012-10-12 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Islet transplant; Kidney transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Subjects with preserved kidney function (Experimental): Subjects with preserved renal function that have not previously received a kidney transplant will be treated with Human Pancreatic Islets (in the form of islets alone - IA).
  Interventions: Drug: Human Pancreatic Islets
- Subjects with prior kidney transplant (Experimental): Subjects with renal failure secondary to diabetes who have received a prior kidney transplant at least 6 months previously and have stable renal function on a steroid-free immunosuppressive regimen will receive Human Pancreatic Islets (in the form of islets after kidney - IAK).
  Interventions: Drug: Human Pancreatic Islets

INTERVENTIONS:
Drug: Human Pancreatic Islets — Pancreatic islet tissue suspended in 150 - 300 ml of phenol red-free CMRL-1066 Transplant Media supplemented with 4% (w/v) HSA and 16mM HEPES in a 600ml transfer pack. Heparin will be administered at 70 IU/kg recipient body weight. Administered by intra-portal vein infusion. To be administered once, however, if full graft function is not achieved, a second or third dose of Pancreatic Islets may be given within 18 months of the first transplant.

SUMMARY:
Islet transplantation can provide physiologic insulin replacement to patients with type 1 diabetes without the complications associated with whole pancreas transplantation. The purpose of this study is to achieve insulin-independence in patients with type 1 diabetes, thereby eliminating the need for exogenous insulin injections to maintain normal glucose levels, ameliorating severe hypoglycemia and potentially decreasing the development of diabetes-related complications. This study will investigate islet transplantation in subjects who have preserved renal function and subjects who have undergone cadaveric renal transplantation, since the latter subjects are already on immunosuppression.

This is a single center, prospective trial of islet transplantation in subjects receiving islets alone or islets after kidney transplant. This is a phase I study investigating the use of islet transplantation for the treatment of type 1 diabetes. Subjects will be eligible for an islet transplant if they meet all of the inclusion criteria and none of the exclusion criteria outlined in the protocol. In brief, the aims of this study are to establish an islet transplant program at the Ohio State University, determine the safety of islet transplantation in islet alone and kidney transplant recipients, determine whether islet transplantation will reduce the frequency of severe hypoglycemic events, determine whether a novel steroid-free immunosuppressive protocol will prevent rejection in islet transplants and to achieve insulin independence at one year after the final islet transplant.

DETAILED DESCRIPTION:
Hypothesis - Insulin independence (insulin injections no longer needed) will be achieved in subjects with type 1 diabetes receiving islet transplantation using the immunosuppressive regimen of cyclosporine and sirolimus. Amelioration of severe hypoglycemia will also be achieved in these groups.

Primary Objective

To determine the safety of islet transplantation in islet alone and in kidney transplant recipients. Safety analyses include:

* Incidence, timing and severity of adverse events and their relationship to the transplant protocol, islet infusion and immunosuppressive medications
* Proportion without protocol-related serious adverse events (SAE) at 1 year
* Incidence, type and severity of infectious complications
* Incidence and severity of procedural-related events, such as bleeding and portal vein thrombosis
* Incidence and severity of liver function test elevations
* Incidence and severity of hypoglycemia
* Incidence and severity of creatinine clearance and urine microalbumin changes
* Incidence and severity of lipid abnormalities
* Proportion of those who develop donor-specific alloantibody

Secondary Objective

To determine the efficacy of islet transplantation in islet alone and in kidney transplant recipients. Efficacy analyses include:

* Time to insulin independence, defined as freedom from insulin use (insulin injections not needed) for 14 or more consecutive days
* Proportion of those that achieve insulin independence at any time during the first year
* Proportion of those one year after final transplant who have:

  * Positive C-peptide (≥0.3 ng/ml after stimulation)
  * Full function of their graft
  * Partial function of their graft
  * Marginal function of their graft
  * Mixed meal stimulated C-peptide >1.0 ng/ml at 6, and 12 months
* Proportion of those that have an acute insulin response to glucose (AIRg) >20uU/ml during frequently sampled intravenous glucose tolerance test (FSIGT) at 6 and 12 months
* Proportion of those with blood glucose level <140 mg/dl two hours after oral glucose tolerance test (OGTT) at 6 and 12 months
* Proportion of those that have improved QOL at 6 and 12 months compared with baseline
* Proportion of those that have improved hypoglycemia and glycemic lability scores at 6 and 12 months compared with baseline

Definition of full islet function:

* Insulin independence
* A1C ≤ 6.5%
* Absence of severe hypoglycemic episodes
* Fasting glucose ≥140 mg/dl less than 3 times a week
* Post-prandial glucose (2 hours) >180 mg/dl less than 4 times a week

Definition of partial islet function:

* Insulin requirement less than 50% of pre-transplant insulin requirement
* C-peptide positive (≥0.3 ng/ml after stimulation)
* A1C ≤ 6.5%
* No severe hypoglycemia

Definition of marginal islet function:

* C-peptide positive (≥0.3 ng/ml after stimulation)
* A1C ≤ 7.5%
* No severe hypoglycemia

This trial will have two study groups consisting of N=10 subjects with type 1 diabetes. One group (IA) will include subjects with preserved kidney function. A second group (IAK) will include subjects with renal failure secondary to diabetes who have received a prior kidney transplant at least 6 months previously and have stable renal function on a steroid-free immunosuppressive regimen.

Potential study participants will be recruited from the Endocrinology and Transplant clinics at the Ohio State University, and community physician referrals. Those who are potentially eligible will undergo a screening evaluation after review of the medical records. If the subject remains eligible, he/she will be enrolled in the islet transplant study and will be placed on a waiting list for an islet transplant. Once a transplant becomes available, the subject will be admitted to the hospital to undergo the transplant procedure. Frequent follow-up visits in the transplant clinic will occur throughout the following year after the transplant. Subjects will be closely monitored for adverse events and insulin requirements. If the subject does not achieve insulin independence, he/she may be eligible for a subsequent transplant.

There will be a 10-year enrollment with 12-month follow-up after last transplant. Since subjects may be eligible for a subsequent transplant within 18 months of the first transplant, the total duration may be up to 30 months after the first transplant in some subjects.

The study will be completed one year after the last islet transplant. Subjects who have undergone the islet transplant procedure and have completed the post-transplant evaluations one year after their last transplant will be considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes > 5 years
2. First islet transplant
3. Demonstrate intensive efforts to manage diabetes for last 6 months (≥4 SMBG/day, ≥3 injections of insulin/day or use of pump and ≥3 contacts with diabetes care team in last 12 months)
4. Metabolic complications: at least one of the following:

   •Reduced hypoglycemia awareness (inability to sense hypoglycemia until blood glucose falls to < 54 mg/dl or > one hypoglycemic episode in last 12 months requiring outside help and not explained by clear precipitant)

   •≥2 severe hypoglycemic events or ≥2 hospitalizations for diabetic ketoacidosis (DKA) in last year.
5. Ability to provide written informed consent
6. Age 18-65
7. Specific for group 2: All of above (1-6) with renal transplant at least 6 months previous

Exclusion Criteria:

1. Age < 18 years or > 65 years
2. Inability to provide informed consent
3. Body Mass Index > 29 kg/m2
4. Insulin requirement of > 50 units/day
5. Stimulated C-peptide ≥ 0.2 ng/ml
6. Current panel reactive anti-HLA antibodies >20%
7. Cardiovascular instability
8. Previous islet transplant
9. History of malignancy except squamous and basal cell skin cancer unless disease-free for > 2 years determined by independent oncologist
10. Active peptic ulcer disease
11. Condition that may interfere with absorption of medications
12. Hemoglobin A1C > 12%
13. Invasive aspergillus infection within one year
14. Varicella titer index <1.0
15. Rubella titer <10 IU/ml
16. Psychiatric disorder
17. Untreated hyperlipidemia: fasting total cholesterol >240 mg/dl, low density lipoprotein>130 mg/dl, or triglycerides >200 mg/dl
18. Hemoglobin <10 g/dl for females, and <11 g/dl for males, white blood cell count < 3,000/µL, platelet count of <150,000/microliter, CD4+ count <500/microliter
19. Liver function test abnormalities (if any value > 1.5 times normal, candidate will be excluded. If 1-1.5 times normal, test will be repeated. If re-test value remains above normal, candidate will be excluded).
20. Prostate specific antigen >4.0 ng/ml
21. Presence of gallstones, liver hemangioma, cirrhosis or evidence of portal hypertension
22. Untreated proliferative diabetic retinopathy
23. Females: positive pregnancy test, intent for future pregnancy, or any subject of reproductive age who is not surgically sterile and is unable or unwilling to use acceptable method of contraception
24. Female subjects who are breast-feeding
25. Adrenal insufficiency: 8am cortisol >19 mcg/dl adequate. Values 19 mcg/dl will be followed by Adreno-Corticotropic Hormone stimulation test
26. Any disease or condition that requires use of chronic steroids
27. Coagulopathy or use of chronic anticoagulation
28. Hyperthyroidism unless treated with radioactive iodine or surgery
29. Thyroid function tests outside normal range
30. Active alcoholism or other substance abuse within the past six months
31. History of non-adherence. Questionable adherence requires agreement entered and compliance demonstrated for at least 3 months
32. Active infection including hepatitis B or C, human immunodeficiency virus positive, positive Mantoux test [unless previously immunized with Bacillus Calmette-Guerin], or X-ray evidence of pulmonary infection
33. Inability to reach hospital within 6 hours of notification
34. Failure to clear psychological or psychiatric screen
35. Medical condition or circumstance that investigator finds will interfere with safe completion of the study

Exclusion criteria specific for group 1:

1. Receipt of previous transplant (excluding pancreas)
2. Creatinine clearance <50 ml/minute for females and <60 ml/minute for males or macroalbuminuria (>500 mg/24h)

Exclusion criteria specific for group 2:

1. Creatinine clearance <40ml/minute
2. Renal transplant in last 6 months
3. Current use of corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
Incidence of serious adverse events | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
  Serious adverse events will be defined (in accordance with FDA Title 21 CFR 312.32) as the following:
  * Death
  * Life-threatening and placing the subject at immediate risk of death
  * Hospitalization
  * Persistent or significant disability or incapacity
  * Congenital abnormal/birth defects
  * Requiring medical or surgical intervention to prevent permanent damage
Incidence of infectious complications | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
Incidence of procedural-related events | Day 1 post-transplant
  Ex. Bleeding or portal vein thrombosis
Incidence of elevated liver function tests | Day 1 post-transplant
Incidence of hypoglycemia | Day 1 post-transplant
Incidence of procedural-related events | Day 2 post-transplant
  Ex. Bleeding or portal vein thrombosis
Incidence of elevated liver function tests | Day 2 post-transplant
Incidence of hypoglycemia | Day 2 post-transplant
Incidence of procedural-related events | Day 3 post-transplant
  Ex. Bleeding or portal vein thrombosis
Incidence of elevated liver function tests | Day 3 post-transplant
Incidence of hypoglycemia | Day 3 post-transplant
Incidence of elevated liver function tests | Day 5 post-transplant
Incidence of hypoglycemia | Day 5 post-transplant
Incidence of elevated liver function tests | Day 7 post-transplant
Incidence of hypoglycemia | Day 7 post-transplant
Incidence of elevated liver function tests | Day 10 post-transplant
Incidence of hypoglycemia | Day 10 post-transplant
Incidence of elevated liver function tests | Day 14 post-transplant
Incidence of hypoglycemia | Day 14 post-transplant
Incidence of elevated liver function tests | Day 21 post-transplant
Incidence of hypoglycemia | Day 21 post-transplant
Incidence of abnormalities in lipids | Day 28 post-transplant
Incidence of elevated liver function tests | Day 28 post-transplant
Incidence of donor-specific antibody development | Day 28 post-transplant
Incidence of hypoglycemia | Day 28 post-transplant
Incidence of elevated liver function tests | Day 42 post-transplant
Incidence of hypoglycemia | Day 42 post-transplant
Incidence of elevated liver function tests | Day 56 post-transplant
Incidence of hypoglycemia | Day 56 post-transplant
Incidence of elevated liver function tests | Day 90 post-transplant
Incidence of hypoglycemia | Day 90 post-transplant
Incidence of abnormalities in lipids | Day 90 post-transplant
Incidence of donor-specific antibody development | Day 90 post-transplant
Incidence of elevated liver function tests | Day 120 post-transplant
Incidence of hypoglycemia | Day 120 post-transplant
Incidence of elevated liver function tests | Day 180 post-transplant
Incidence of hypoglycemia | Day 180 post-transplant
Incidence of abnormalities in lipids | Day 180 post-transplant
Incidence of donor-specific antibody development | Day 180 post-transplant
Incidence of elevated liver function tests | Day 270 post-transplant
Incidence of hypoglycemia | Day 270 post-transplant
Incidence of abnormalities in lipids | Day 270 post-transplant
Incidence of donor-specific antibody development | Day 270 post-transplant
Incidence of elevated liver function tests | Day 365 post-transplant
Incidence of abnormalities in lipids | Day 365 post-transplant
Incidence of hypoglycemia | Day 365 post-transplant
Incidence of donor-specific antibody development | Day 365 post-transplant
Change in microalbumin level | Days 180 and 365 post-transplant
Change in measured creatinine clearance | Days 180 and 365 post-transplant

SECONDARY OUTCOMES:
Amount of daily insulin units required | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
Measurement of C-peptide | Days 1, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
Change in c-peptide level from fasting following administration of mixed meal | Days 180 and 365 post-transplant
  Patients fasting c-peptide will be measured, then patient will be given a mixed meal of Ensure. The c-peptide level will be checked again at 90 minutes after administration of mixed meal.
Change in acute insulin response to glucose | Days 180 and 365 post-transplant
  As determined by oral glucose tolerance test and/or intravenous glucose tolerance test
Incidence of blood glucose level <140mg/dl two hours after oral glucose tolerance tests | Days 180 and 365 post-transplant
Change in Quality of Life | Days 180 and 365 post-transplant
Change in hypoglycemia score | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant
Change in glycemic lability score | Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 90, 120, 180, 270 and 365 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Amer Rajab, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data for patients who agree is entered into a multi-center islet transplant data registry (no personally identifiable information will be shared). Upon completion of the study, results may also be published in a peer-reviewed journal.